CLINICAL TRIAL: NCT00624585
Title: A Pilot Study of Oral Dasatinib in Subjects With MDS and Excess Marrow Blasts
Brief Title: Study of Oral Dasatinib in Subjects With Myelodysplastic Syndrome (MDS) and Excess Marrow Blasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15276; CA180-106 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; MDS/MPD; MDS/AML; CMML; Excess Marrow Blasts
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib Dose Escalation (Experimental): Patients will be started on dasatinib at a continuous oral daily dose of 100 mg per day. At 8 weeks, if the initial dose is well tolerated and patient has not achieved a partial response, the dose may be increased to 150 mg per day. All patients will be followed per protocol for a total core period of 16 weeks from the first dose. Responding patients will continue dasatinib treatment for up to 48 weeks in the absence of treatment failure, disease progression, limiting toxicity or death. Patients continuing after 48 weeks will be enrolled in a separate extension study for future follow up.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — DOSE ESCALATION OF DASATINIB AFTER 8 WEEKS IF ELIGIBLE
  * Dose Level and Dose of dasatinib:
    1. Starting dose (1-8 weeks)= 100 mg orally (po) daily
    2. +1 (<8 weeks if no PR and well tolerated) = 150 mg po daily
  DOSE MODIFICATION OF DASATINIB
  * Dose Level and Dose of dasatinib:
    1. Starting dose = 100 mg po daily
    2. -1 = 70 mg po daily
    3. -2 = 50 mg po daily
  OR
  * Dose Level and Dose of dasatinib:
    1. Starting dose = 150 mg po daily
    2. -1 = 120 mg po daily
    3. -2 = 90 mg po daily
    4. -3 = 50 mg po daily
  Other Names: SPRYCEL®

SUMMARY:
The main purpose of this study is to learn how patients with myelodysplastic syndrome (MDS) respond to the study drug dasatinib. The study drug, dasatinib, has been approved by the U.S. Food and Drug Administration (FDA) for treatment of leukemia, but has not been approved for the treatment of other kinds of cancer. The use of dasatinib in this study is considered experimental.

DETAILED DESCRIPTION:
Study Core Period:

The first 16 weeks after the initial dose of dasatinib is called the Study Core Period. Patients who are eligible and chose to participate in this study should expect to take 100 mg of dasatinib daily for 8 weeks. If the study doctor believes that they have not achieved a partial response after 8 weeks of treatment, the dose may be increased to 150 mg per day. The study doctor may lower the dosage of dasatinib if the 100 mg treatment is too strong. If the lower dose of dasatinib is still too strong, the study doctor may decide to take the patient off of the study. The patient will continue to receive supportive care as needed during the duration of the trial as well as after completion of the trial.

During the Study Core Period, participants will have a study visit every 4 weeks. Complete Blood Counts (CBCs) will be obtained every 2 weeks for study purposes and disease monitoring. Bone marrow aspiration and biopsy will be obtained at screening, and at 8 weeks and 16 weeks of treatment for response assessment. Additional bone marrow aspirations and biopsies may be obtained at any other time, to evaluate the disease process, at the doctor's judgment. A bone marrow aspirate and biopsy must be done at the time of study discontinuation.

Study Extension Period:

The time after the first 16 weeks of treatment is called the study extension period. If the patient is responding to the treatment, does not experience disease progression or any severe adverse events, the patient may continue dasatinib treatment for up to 48 weeks. If patients continue after 48 weeks, they will be asked to enroll in a separate extension study for future follow up.

During the Study Extension Period, participants will have a study visit every 4 weeks. Complete Blood Counts (CBCs) will be obtained every 2 or 4 weeks for study purposes and disease monitoring. Bone marrow aspiration and biopsy will be obtained every 16 weeks. A bone marrow aspirate and biopsy must be done at the time of study discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MDS or Myeloproliferative Disorders (MPS/MPD) with blast percentage > 10% in bone marrow, MDS/AML with <30% blasts:

  * MDS [all World Health Organization (WHO) types] with blast percentage > 10% in bone marrow
  * Chronic myelomonocytic leukemia (CMML) with blast percentage > 10% in bone marrow
  * Myelodysplastic / Myeloproliferative (MDS/MPD) syndromes with blast percentage > 10% in bone marrow
  * Acute myeloid leukemia with Multilineage Dysplasia (MDS/AML) with <30% blasts and declined standard induction chemotherapy or deemed unfit for standard induction chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
* Previous therapy with Azacitidine or Decitabine with last dose at least 2 months prior to first dose of dasatinib okay. Must be at least 4 weeks out from any previous investigational therapy.
* Adequate Organ Function

  * Total bilirubin < 2.0 times institutional Upper Limit of Normal (ULN)
  * Hepatic enzymes (AST, ALT) ≤ 2.5 times institutional ULN
  * Serum Na, K+, Mg2+, Phosphate and Ca2+≥ Lower Limit of Normal (LLN) [low electrolyte levels must be repleted to all for entry]
  * Serum Creatinine < 1.5 times ULN
  * Prothrombin time (PT), partial thromboplastin time (PTT) Grade 0-1
* Able to take oral medication (Dasatinib must be swallowed whole. Tablets can be dissolved in juice and then put down an NG/G tube or drank as a solution)
* Women of childbearing potential (WOCBP) must have Negative serum or urine pregnancy test within 72 hours prior to start of study drug
* Persons of reproductive potential must agree to use adequate birth control throughout treatment and at least 4 weeks after study drug is stopped
* Signed written informed consent

Exclusion Criteria:

* White blood count (WBC) >50,000 off hydroxyurea for >72 hours
* Malignancy [other than the one treated in this study] requiring radiotherapy or systemic treatment within past 3 years
* Chemotherapy or any agent with activity in MDS or AML concurrent with the study.
* Chemotherapy for MDS or AML prior to enrollment not allowed other than Azacitidine or Decitabine >2 months prior to first dose
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Pleural or pericardial effusion
  * Serious medical condition, unstable medical co-morbidity, psychiatric illness that will prevent subject from signing informed consent form or place them at unacceptable risk if they participate
* Cardiac Symptoms, including:

  * Uncontrolled angina, congestive heart failure or myocardial infarction (MI) within 6 months
  * Diagnosed congenital long QT syndrome
  * History of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes)
  * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Hypokalemia or hypomagnesemia if cannot be corrected
* History of significant bleeding disorder unrelated to cancer, including:

  * Congenital bleeding disorders
  * Acquired bleeding disorder within 1 year
  * Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding
* Concomitant Medications, consider the following prohibitions:

  * Drugs generally accepted to have risk of causing Torsades de Pointes(Must discontinue drug 7 days prior to starting dasatinib)
  * Concomitant use of H2 blockers or proton pump inhibitors with dasatinib not recommended. Use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy.
  * On-going requirement for treatment with platelet function inhibitor or anti-coagulation.
  * Must discontinue St. Johns Wort while receiving dasatinib therapy
  * Must agree that intravenous (IV) bisphosphonates be withheld for first 8 weeks of Dasatinib therapy due to risk of hypocalcemia.
  * May not be receiving any prohibited CYP3A4 inhibitors
* Women:

  * Positive pregnancy test at baseline
  * Pregnant or breastfeeding
* Prisoners or patients who are compulsorily detained for treatment of either psychiatric or physical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan List, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Int-2 or High risk MDS according to International Prognostic Scoring System (IPSS) score. All World Health Organization (WHO) subtypes of Myelodysplastic Syndrome (MDS), Chronic Myelomonocytic Leukemia (CMML), or Myelodysplastic / Myeloproliferative (MDS/MPD) were allowed.
Pre-assignment Details: Acute Myeloid Leukemia Multilineage Dysplasia (MDS/AML) with <30% blasts (RAEB-t) who either declined or were deemed unfit for induction chemotherapy were also eligible. Exclusion criteria were WBC >50,000 off hydroxyurea, another malignancy requiring radiation or chemotherapy within the past 3 years, or concurrent therapy for MDS or AML.
Groups:
- Dasatinib Dose Escalation: Patients were started on dasatinib at a continuous oral daily dose of 100 mg per day. At 8 weeks, if the initial dose was well tolerated and patient had not achieved a partial response, the dose could be increased to 150 mg per day. All patients were followed per protocol for a total core period of 16 weeks from the first dose. Responding patients could continue dasatinib treatment for up to 48 weeks in the absence of treatment failure, disease progression, limiting toxicity or death. Patients continuing after 48 weeks will be enrolled in a separate extension study for future follow up.
Period: Overall Study
Arm/Group | Dasatinib Dose Escalation
Started | 18
Completed | 6
Not Completed | 12
Not completed — Death | 3
Not completed — Disease Progression | 6
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib Dose Escalation
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [60 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Marrow Complete Remission (CR)
Description: Complete remission (modified IWG); IWG = International MDS Working Group.
  Bone Marrow Response must last ≥4 weeks. Bone marrow evaluation: Bone marrow showing ≤5% myeloblasts with normal maturation of all cell lines.
Time Frame: 1 Year 4 Months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Dasatinib Dose Escalation
Number analyzed (Participants) | 18
participants | 3

2. Secondary Outcome: Number of Participants With Hematologic Improvement
Description: Hematologic improvement in platelets, red blood cell (RBC), neutrophils according to modified IWG Criteria; Cytogenetic response (modified IWG); Change in percentage of blasts in bone marrow and peripheral blood; Src-Tyr416 phosphorylation in medullary myeloblasts. Hematologic improvements must last ≥ 8 weeks.
Time Frame: 1 Year 4 Months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Dasatinib Dose Escalation
Number analyzed (Participants) | 18
participants | 0

3. Secondary Outcome: Number of Participants With Partial Remission (PR)
Description: Partial remission (PR) (modified IWG); IWG = International MDS Working Group. All of the CR criteria (if abnormal prior to treatment), except: Bone marrow evaluation: Blasts decreased by ≥ 50% over pretreatment but still >5%. Cellularity and morphology are not relevant.
Time Frame: 1 Year 4 Months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Dasatinib Dose Escalation
Number analyzed (Participants) | 18
participants | 0

4. Secondary Outcome: Number of Participants With Stable Disease (SD)
Time Frame: 1 Year 4 Months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Dasatinib Dose Escalation
Number analyzed (Participants) | 18
participants | 10

ADVERSE EVENTS:
Time Frame: 1 Year 4 Months
Arm/Group | Dasatinib Dose Escalation
Serious Adverse Events (participants affected / at risk) | 9/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib Dose Escalation (N=18)
Anorexia - Grade 3 - *Possibly related (Gastrointestinal disorders) | 1 (1)
Blood/Bone Marrow - Grade 4 (Blood and lymphatic system disorders) | 1 (1)
Cardiac general - Grade 3 (Cardiac disorders) | 1 (1)
Cholecystitis - Grade 3 - *Possibly related (Hepatobiliary disorders) | 1 (1)
Confusion - Grade 3 (Nervous system disorders) | 1 (1)
Dehydration - Grade 3 (Gastrointestinal disorders) | 1 (1)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 1 (1)
Diarrhea - Grade 3 - *Possibly related (Gastrointestinal disorders) | 1 (1)
Dyspnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea - Grade 2 - *Possibly related (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea - Grade 3 - **Definitely related (Respiratory, thoracic and mediastinal disorders) | 1 (1) — **"Definitely related to study" events are noted as appropriate
Dyspnea - Grade 3 - *Possibly related (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Edema: limb - Grade 2 (Blood and lymphatic system disorders) | 2 (2)
Fatigue - Grade 3 - *Possibly related (General disorders) | 3 (4)
Febrile neutropenia - Grade 3 (Infections and infestations) | 1 (1)
Febrile neutropenia - Grade 3 - *Possibly related (Infections and infestations) | 1 (1) — *"Possibly related to study" events are noted as appropriate
Fever in absence of neutropenia - Grade 2 (General disorders) | 1 (1)
Glucose, serum - low - Grade 4 (Metabolism and nutrition disorders) | 1 (1)
Hematoma - Grade 1 (General disorders) | 1 (1)
Hemoglobin - Grade 3 - *Possibly related (Blood and lymphatic system disorders) | 3 (4)
Hemoglobin - Grade 4 - *Possibly related (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI - Lower GI NOS - Grade 3 (General disorders) | 1 (1)
Hemorrhage, GI - Rectum - Grade 3 - *Possibly related (General disorders) | 1 (1)
Hemorrhage, GI - Upper GI - Grade 3 - *Possibly related (General disorders) | 1 (1)
Hepatobiliary/Pancreas - Grade 1 (Hepatobiliary disorders) | 1 (1)
Hypertension - Grade 3 (Cardiac disorders) | 1 (1)
Infection - Grade 3 (Infections and infestations) | 2 (2)
Infection - Grade 3 - *Possibly related (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung - Grade 3 (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - lung - Grade 3 - *Possibly related (Infections and infestations) | 1 (1)
Mucositis/stomatitis (oral cavity) - Grade 3 (Gastrointestinal disorders) | 1 (2)
Nausea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 3 - *Possibly related (Gastrointestinal disorders) | 1 (1)
Pain - Cardiac/heart - Grade 3 (General disorders) | 1 (1)
Pain - head/headache - Grade 3 (General disorders) | 1 (1)
Pain: abdomen - Grade 2 (General disorders) | 2 (2)
Platelets - Grade 3 - *Possibly related (Blood and lymphatic system disorders) | 1 (1)
Platelets - Grade 4 - *Possibly related (Blood and lymphatic system disorders) | 2 (2)
Pleural effusion - Grade 2 - **Definitely related (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion - Grade 2 - *Possibly related (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion - Grade 3 - *Possibly related (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure - Grade 3 (Renal and urinary disorders) | 1 (1)
Renal failure - Grade 3 - *Possibly related (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Grade 2 (Renal and urinary disorders) | 1 (1)
Vomiting - Grade 1 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 2 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 3 - *Possibly related (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib Dose Escalation (N=18)
Alergic rhinitis (Immune system disorders) | 1 (1)
Anorexia - *2 Events possibly related (Gastrointestinal disorders) | 3 (3)
Auditory/Ear (Ear and labyrinth disorders) | 1 (1)
Blood/Bone Marrow - *Possibly related (Blood and lymphatic system disorders) | 1 (1) — *"Possibly related to study" events are noted as appropriate
Bruising (in absence of Grade 3 or 4 thrombocytopenia) - *2 Events possibly related (Skin and subcutaneous tissue disorders) | 6 (6)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Cardiac troponia I (cTnl) (Cardiac disorders) | 1 (1)
Constipation - *3 Events possibly related (Gastrointestinal disorders) | 4 (4)
Cough - *3 Events possibly related (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dehydration - *Possibly related (Gastrointestinal disorders) | 1 (1)
Dermatology (Skin and subcutaneous tissue disorders) | 5 (6)
Diarrhea - *5 Events possibly related (Gastrointestinal disorders) | 8 (8)
Dizziness (General disorders) | 1 (1)
Dysgeusia - *4 Events possibly related (Gastrointestinal disorders) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea - *6 Events possibly related (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Edema: limb - *3 Events possbily related (Blood and lymphatic system disorders) | 4 (4)
Fatigue - *13 Events possibly related (General disorders) | 12 (20)
Febrile neutropenia - *3 Events possibly related (Infections and infestations) | 4 (4)
Fever (General disorders) | 1 (1)
Flushing - *Possibly related (Skin and subcutaneous tissue disorders) | 1 (1)
Gastrointestinal - other - *3 Events possibly related (Gastrointestinal disorders) | 5 (9)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (3)
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin - *11 Events possibly related (Blood and lymphatic system disorders) | 6 (12)
Hemorrhage, GI - Oral cavity (General disorders) | 1 (2)
Hemorrhage, GI - Rectum - *1 Event possibly related (General disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory - Lung - *Possibly related (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypoxia - *Possibly related (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - other - *2 Events possibly related (Infections and infestations) | 4 (6)
Infection with Grade 3 or 4 neutrophils - Urinary tract - *Possibly related (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Skin - *Possibly related (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus - *1 Event possibly related (Infections and infestations) | 2 (3)
Insomnia (General disorders) | 2 (2)
Iron overload (Blood and lymphatic system disorders) | 1 (2)
Leukocytes (total WBC) - *Possibly related (Blood and lymphatic system disorders) | 2 (2)
Lymphatics (Blood and lymphatic system disorders) | 2 (2)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Mucositis/stomatitis - Oral cavity - *Possibly related (Gastrointestinal disorders) | 1 (1)
Muscle weakness - *2 Events possibly related (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea - *Possibly related (Gastrointestinal disorders) | 6 (6)
Neuropathy - *Possibly related (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) - *Possibly related (Blood and lymphatic system disorders) | 1 (4)
Ocular/Visual - *1 Event possibly related (Eye disorders) | 4 (4)
Pain (General disorders) | 3 (5)
Pain - Abdomen - *2 Events possibly related (General disorders) | 3 (4)
Pain - Back (General disorders) | 2 (2)
Pain - Breast (General disorders) | 1 (1)
Pain - Chest wall - *1 Event possibly related (General disorders) | 2 (3)
Pain - Extremity: limb (General disorders) | 1 (3)
Pain - Head/headache - *4 Events possibly related (General disorders) | 3 (6)
Pain - Joint - *Possibly related (General disorders) | 1 (2)
Pain - Oral cavity (General disorders) | 2 (2)
Pain - Throat/pharynx/larynx - *1 Event possibly related (General disorders) | 2 (2)
Platelets - *6 Events possibly related (Blood and lymphatic system disorders) | 6 (8)
Pleural effusion - *Possibly related (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Potassium, serum-low (hypokalemia) - *1 Event possibly related (Metabolism and nutrition disorders) | 2 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary/Upper Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation - *Possibly related (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: hand-foot skin reaction - *Possibly related (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure - *Possibly related (Renal and urinary disorders) | 1 (1)
Rigors/chills - *1 Event possibly related (General disorders) | 3 (3)
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) - *1 Event possibly related (General disorders) | 3 (3)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vomiting - *Possibly related (Gastrointestinal disorders) | 1 (2)
Weight loss - *Possibly related (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes